CLINICAL TRIAL: NCT01930240
Title: A Randomized Placebo Controlled Double Blind Two Period Cross-Over Study to Assess the Safety and Pharmacokinetics and Pharmacodynamics of Oral Dosages of TRIA-662 (A Hypolipidemic Agent) in Healthy Volunteers
Brief Title: The Safety of a Hypolipidemic Agent in Healthy Normal Volunteers
Acronym: Cortria-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortria Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Cortria-002
Record Dates: First submitted 2013-08-21; First posted 2013-08-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TRIA-662 Placebo (Placebo Comparator): Single dose of nine placebo capsules matching TRIA-662 drug capsules
  Interventions: Drug: Placebo
- TRIA-662 Low Dose (Experimental): Single-dose of TRIA-662 administered as three 30 mg TRIA-662 capsules and six matching placebo capsules
  Interventions: Drug: TRIA-662
- TRIA-662 High Dose (Experimental): Single dose of TRIA-662 administered as nine 30mg TRIA-662 capsules
  Interventions: Drug: TRIA-662

INTERVENTIONS:
Drug: TRIA-662 — 1-MNA Chloride
  Other Names: 1-MNA Chloride
  Arms: TRIA-662 High Dose; TRIA-662 Low Dose
Drug: Placebo — Double-blind placebo
  Other Names: Dummy
  Arms: TRIA-662 Placebo

SUMMARY:
The primary objective of the study is to assess the blood profile of the N-methylnicotinamide (MNA) following administration of TRIA-662 (N-methylnicotinamide Chloride). The secondary objectives of the study are to characterize the safety and tolerability of TRIA-662 and to assess any potential gender-related differences in the plasma profile of MNA. Changes in serum lipid parameters with particular reference to triglycerides, lipoprotein lipase, and blood pressure effects will also be noted.

DETAILED DESCRIPTION:
A total of 20 subjects volunteers (10 male and 10 female) will receive the following treatments administered in a randomized fashion with 2 embedded placebo dosages in each group (8 active Males and 8 active females with 2 placebo males and females):

1. DRUG (Low Dose): Single therapeutic dose of MNA administered as a 90 mg oral dose
2. DRUG (High Dose): Single therapeutic dose of MNA administered as a 270 mg oral dose
3. PLACEBO: Placebo for MNA administered as an identically appearing oral dose Each treatment period will consist of a 3-day two-night confinement cycle with admission on day 1, treatment on day 1 with a single dose of active or placebo with discharge 24 hours following the last assessment the next morning. A washout period of 5 days will separate each treatment period. Standard biochemical and clinical baseline medical background and physical examination will occur at screening and at Day -1 to assess/confirm entry criteria. During each treatment period, serial plasma samples (n=12) for MNA assay will be collected on the treatment day. Safety assessments, including vitals signs (blood pressure, pulse rate, respiration rate, and oral body temperature), will be performed at screening, at baseline, and at 4 times throughout each treatment period. Physical examinations and standard clinical laboratory tests (hematology, serum chemistry, and urinalysis) will be obtained at screening, and at admission for each treatment period, and prior to subject's final discharge from the study. The Lunch meals on the dosing day will be identical in each subject on each occasion.

The pharmacokinetic and safety assessments will be performed at specified times prior to and after study MNA administration.

ELIGIBILITY:
Inclusion Criteria:

1. Good health (based on medical history, physical examination, electrocardiogram, and clinical laboratory tests)
2. Non-smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the Screening visit)
3. Between 18 and 50 years old (inclusive)
4. Body weight within 20% of the desirable weight for adults at the Screening visit
5. Able to execute informed written consent (informed consent must be obtained for all subjects before enrollment in the study.
6. Willingness to abstain from alcohol and xanthine-containing food and beverages for the duration of each treatment period
7. Willingness to remain in the clinic for the inpatient portions of the study
8. Female subjects must be non-pregnant and either surgically sterile, postmenopausal for a least 1 year, or using an acceptable method of contraception defined as an oral, implanted, or transdermal contraceptive plus one of the following barrier methods: diaphragm with spermicidal cream/jelly or use of a condom by sexual partner.

Exclusion Criteria:

1. Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years
2. Unwilling or unable to comply with the protocol or reside in the study unit during the study period or to cooperate fully with the principal investigator and site personnel
3. Has used any 1) prescription medication within 14 days prior to treatment in either treatment period or 2), or any over-the-counter (OTC) medication, herbal preparations, and/or vitamins within 48 hours prior to the start of study MNA administration on either treatment period of this study.
4. Has a clinically abnormal ECG
5. Has a serum potassium, sodium, calcium, or magnesium level that is not within normal limits or has other vital signs or clinical laboratory values at the screening visit that are deemed by the principal investigator to make the subject an inappropriate candidate for the study
6. Has taken any other investigational drug during the 30 days prior to screening visit
7. Has donated or lost more than a unit of blood within 30 days prior to screening visit
8. History of renal, hepatic, gastrointestinal, cardiovascular, or hematologic disease
9. Serious mental or physical illness within the past year
10. Has any condition(s) that in the investigator's opinion would: a) warrant exclusion from the study or b) prevent the subject from completing the study
11. Have a positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody at screening
12. Be a female subject with a positive serum pregnancy test or who is breast-feeding at screening
13. Be unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available
14. Has a history of hypersensitivity or allergic reaction to Niacin or Nicotinamide
15. Has had prior exposure to MNA
16. Has a Mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the side effects or tolerance of the study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
MNA Maximum plasma concentration (Cmax). | 0, 1, 2, 3, 4, 5, 8, 12, 18, 24 hours after dose.
  5 mL venous blood samples will be collected by venipuncture at the specified times. These blood samples will be properly processed and analyzed for concentration of MNA and metabolites. The concentration data will undergo typical pharmacokinetic data analysis to arrive at the primary endpoints.
Time to plasma MNA Cmax | 0, 1, 2, 3, 4, 5, 8, 12, 18, 24 hours after dose.
  5 mL venous blood samples will be collected by venipuncture at the specified times. These blood samples will be properly processed and analyzed for concentration of MNA and metabolites. The concentration data will undergo typical pharmacokinetic data analysis to arrive at the primary endpoints.
Area under the plasma MNA concentration curve | 0, 1, 2, 3, 4, 5, 8, 12, 18, 24 hours after dose.
  5 mL venous blood samples will be collected by venipuncture at the specified times. These blood samples will be properly processed and analyzed for concentration of MNA and metabolites. The concentration data will undergo typical pharmacokinetic data analysis to arrive at the primary endpoints.

IPD SHARING:
Plan to Share IPD: No